CLINICAL TRIAL: NCT01676974
Title: Impact of International Travel on the Emergence and Spread of Antimicrobial Resistance in The Netherlands
Brief Title: Carriage Of Multiresistant Bacteria After Travel
Acronym: COMBAT
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Maastricht University Medical Center (Other); Erasmus Medical Center (Other); Utrecht University (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Menno D. de Jong, MD, Prof. dr. M.D. de Jong, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: COMBAT
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Enterobacteriaceae, Infection
Keywords: Drug Resistance, Microbial; Enterobacteriaceae; ESBL; Carbapenemase; Travel
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal Swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Travelers: Travelers and their family members

SUMMARY:
Objectives: Prospectively study the influence of foreign travel and associated risk factors on the acquisition of AMR in the endogenous microbiota of healthy individuals and the subsequent persistence of AMR carriage and transmission to household members of these carriers. Examine whether carriers of resistant Enterobacteriaceae have a higher risk of bacterial infections in the year after travel (compared to non-carriers). Explore the full width of AMR genes and transferable genetic elements acquired during international travel.

DETAILED DESCRIPTION:
Rationale: Antimicrobial resistance (AMR) among Enterobacteriaceae constitutes an increasingly important human health hazard worldwide. Also in the Netherlands AMR rates have been on the rise in recent years. A limited number of previous studies have suggested high acquisition rates of AMR E. coli during international travel, but information on travel-associated risk factors, duration of colonization and local transmission of imported AMR are largely, if not entirely, lacking.

Objectives: Prospectively study the influence of foreign travel and associated risk factors on the acquisition of AMR in the endogenous microbiota of healthy individuals and the subsequent persistence of AMR carriage and transmission to household members of these carriers. Examine whether carriers of resistant Enterobacteriaceae have a higher risk of bacterial infections in the year after travel (compared to non-carriers). Explore the full width of AMR genes and transferable genetic elements acquired during international travel.

Study design: multicenter longitudinal cohort study.

Study population: healthy, adult (> 18 years) volunteers travelling abroad for 1 week - 3 months. Non travelling household members of these traveling volunteers.

Methods: Travelers and non-traveling household members will be recruited at outpatient travel clinics throughout The Netherlands. Faecal samples and questionnaires will be taken before (t=0) travel, immediately after travel (t=1) and 1 month upon return (t = 2). For volunteers that acquire AMR Enterobacteriaceae, repeated questionnaires and faecal samples will be taken after 3, 6 and 12 months.

Faecal samples will be cultured to screen for AMR Enterobacteriaceae. Suspected colonies will be identified and susceptibilities confirmed by standard methods. Genotypic characterization of the extended-spectrum betalactamase- (ESBL-) and carbapenemase genes will be performed using microarray and gene sequencing. Clonal bacterial spread within households will be confirmed or excluded by molecular typing.

Outcomes: The main outcome measure is the acquisition rate and persistence of AMR in the endogenous microbiota of healthy travelers upon travel.

Secondary outcomes are the duration of colonization, the rate of secondary transmission within households, the identification of risk factors, occurrence of self-reported infections in the year following travel and the abundance and type of resistance.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* travelling for > 1 week (7 days) AND < 3 months (90 days)
* non traveling household members of these traveling volunteers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Travelers and their family members not planning to travel
Sampling Method: Probability Sample
Enrollment: 2215 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
acquisition rate | 1 year
  the acquisition rate and persistence of AMR in the endogenous microbiota of healthy travelers upon travel

SECONDARY OUTCOMES:
duration of colonization | 1 year
rate of secondary transmission within households | 1 year
identification of risk factors | 1 year
occurrence of self-reported infections in the year following travel | 1 year
abundance and type of resistance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Menno D. de Jong, PhD, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (3):
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Erasmus Medisch Centrum, Rotterdam

REFERENCES:
- [Derived] Arcilla MS, van Hattem JM, Haverkate MR, Bootsma MCJ, van Genderen PJJ, Goorhuis A, Grobusch MP, Lashof AMO, Molhoek N, Schultsz C, Stobberingh EE, Verbrugh HA, de Jong MD, Melles DC, Penders J. Import and spread of extended-spectrum beta-lactamase-producing Enterobacteriaceae by international travellers (COMBAT study): a prospective, multicentre cohort study. Lancet Infect Dis. 2017 Jan;17(1):78-85. doi: 10.1016/S1473-3099(16)30319-X. Epub 2016 Oct 14. PMID 27751772
- [Derived] Arcilla MS, van Hattem JM, Bootsma MC, van Genderen PJ, Goorhuis A, Schultsz C, Stobberingh EE, Verbrugh HA, de Jong MD, Melles DC, Penders J. The Carriage Of Multiresistant Bacteria After Travel (COMBAT) prospective cohort study: methodology and design. BMC Public Health. 2014 Apr 28;14:410. doi: 10.1186/1471-2458-14-410. PMID 24775515